CLINICAL TRIAL: NCT03907345
Title: Generalized Fear Extinction to Untreated Fear Stimuli in Specific Phobias After Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Armin Zlomuzica, Principal Investigator, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AZ 032019
Record Dates: First submitted 2019-03-28; First posted 2019-04-08 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Fear of Spiders; Fear of Heights
Keywords: Exposure Therapy; Fear of Spiders; Fear of Heights; Anxiety Disorders; Generalization; Extinction; Specific Phobias
MeSH Terms: conditions — Arachnophobia; Acrophobia; Anxiety Disorders; Phobia, Specific

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure (Experimental): Participants of this arm receive one 120-minute session of exposure treatment for spider fear.
  Interventions: Behavioral: Exposure
- No Exposure (No Intervention): Participants of this arm receive no exposure or other adequate treatment.

INTERVENTIONS:
Behavioral: Exposure — The exposure session comprises a hierarchy of 7 steps, reaching from (1) holding a glass with the spider 30cm in from the body / face, to (7) letting the spider walk on the arm. The exposure session has a duration of 120 minutes. Prior to the exposure, participants receive psychoeducation on anxiety and phobias. A house spider (Tegenaria domestica) is used for the exposure.
  Arms: Exposure

SUMMARY:
This study investigates whether a one-session exposure treatment for spider-related stimuli can lead to a generalization of extinguished fear to height-related stimuli in individuals with comorbid fear of spiders and fear of heights.

DETAILED DESCRIPTION:
Exposure therapy has been proven to be effective in the treatment of specific phobias and in a variety of fear evoking situations and stimuli. However, since there is a high prevalence of comorbid fears, therapeutic interventions can get very extensive when each fearful situation and / or stimuli needs to be treated separately and over a repeated number of times. It has recently been shown, that exposure to one fearful stimuli (i.e., a spider), can also lead to a reduction of fear to another, perceptually and conceptually related, but untreated fearful stimulus (i.e., a cockroach) (Preusser, Margraf & Zlomuzica, 2017). Potentially, this generalization of exposure effects might also be relevant for coexisting fears that do not share conceptually related fearful stimuli (e.g., fear of spiders and fear of heights). The present study aims to investigate whether successful exposure treatment to one fearful stimulus (i.e., a spider) can also lead to a reduction of fear to an untreated fear evoking stimulus (i.e., height).

Participants will be randomly assigned to the treatment or no-treatment condition. The entire experimental procedure will take place in three sessions. The first session incorporates spider and height fear related questionnaires and two Behavioral Approach Tests (BATs): One that involves a spider and one that involves height. These BATs are counterbalanced in each group with half of participants receiving the spider BAT first and the height BAT second, and vice versa. The second session takes place approximately seven days later. The treatment group receives a seven-step in vivo exposure with spiders (duration: 1,5 hours). Twenty-four hours later, session 3 takes place and involves the same measures that were applied in session 1. The treatment and no-treatment group receive an identical set of measures except that the no-treatment group will not be subjected to exposure. The effects of exposure-based anxiety reductions toward spiders (treated fear stimulus) and heights (untreated fear stimulus to assess generalization of treatment outcome) are assessed on the behavioral and subjective level at pretreatment and posttreatment (24 hours after exposure).

ELIGIBILITY:
Inclusion Criteria:

* Comorbid presence of fear of spiders and fear of heights [Potential diagnosis of specific phobias (arachnophobia and acrophobia) assessed by application of the Diagnostic Short-Interview for Mental Disorders (Mini-Dips)].

Exclusion Criteria:

* Any acute or chronic mental and / or somatic disease
* Psychological, psychiatric, neurological or pharmacological treatment (Application of the Mini-DIPS to screen for the presence of a psychological condition)
* Drug or alcohol abuse
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Behavioral Approach Test (BAT) for Spiders | Change in BAT scores from pre- to posttreatment (across one week from pretreatment to posttreatment)
  Change in the Behavioral Approach Test (BAT) with spiders (treated fear stimulus) [Time Frame: Pretreatment (approx. 1 week before the treatment), Posttreatment (1 day after treatment), Follow-up (4 weeks between treatment and follow-up)].
  During the Behavioral Approach Test (BAT) the closest distance to a spider as well as subjective fear and heart rate is measured.
Behavioral Approach Test (BAT) for Heights | Change in BAT scores from pre- to posttreatment (across one week from pretreatment to posttreatment)
  Change in the Behavioral Approach Test with heights (untreated fear stimulus) [Time Frame: Pretreatment (approx. 1 week before the treatment), Posttreatment (1 day after treatment), Follow-up (4 weeks between treatment and follow-up)].
  During the Behavioral Approach Test (BAT) the level of the approached height as well as subjective fear and heart rate is measured.

SECONDARY OUTCOMES:
Fear of Spiders Questionnaire (FSQ) | Change in FSQ scores from pre- to posttreatment (across one week from pretreatment to posttreatment)
  Change in the Spider-fear related questionnaires [Time Frame: Pretreatment (approx. 1 week before the treatment), Posttreatment (1 day after treatment), Follow-up (4 weeks between treatment and follow-up)].
  Self-report questionnaires assessing fear of spiders will be used. The Fear of Spiders Questionnaire (FSQ) will be applied. Scores on this scale range from 0 to 108, with higher scores indicating greater fear of spiders.
Spider Fear Questionnaire (SPQ) | Change in SPQ scores from pre- to posttreatment (across one week from pretreatment to posttreatment)
  Change in the Spider-fear related questionnaires [Time Frame: Pretreatment (approx. 1 week before the treatment), Posttreatment (1 day after treatment), Follow-up (4 weeks between treatment and follow-up)].
  Self-report questionnaires assessing fear of spiders will be used. The Spider Fear Questionnaire (SPQ) will be applied. Scores on this scale range from 0 to 31, with higher scores indicating greater fear of spiders.
Spider Beliefs Questionnaire (SBQ) | Change in SBQ scores from pre- to posttreatment (across one week from pretreatment to posttreatment)
  Change in the Spider-fear related questionnaires [Time Frame: Pretreatment (approx. 1 week before the treatment), Posttreatment (1 day after treatment), Follow-up (4 weeks between treatment and follow-up)].
  Self-report questionnaires assessing fear of spiders will be used. The Spider Beliefs Questionnaire (SBQ) will be applied. Scores on this scale range from 0 to 100, with higher scores indicating greater fear of spiders.
Acrophobia Questionnaire (AQ) | Change in AQ scores from pre- to posttreatment (across one week from pretreatment to posttreatment)
  Change in the height related questionnaire [Time Frame: Pretreatment (approx. 1 week before the treatment), Posttreatment (1 day after treatment), Follow-up (4 weeks between treatment and follow-up)].
  Self-report questionnaires assessing fear of heights will be used. The German version of the anxiety subscale of the Acrophobia Questionnaire (AQ) will be used. Scores on these scales range from 0 to 120, with higher scores indicating greater fear of heights.

OTHER OUTCOMES:
Fear and Disgust Rating | Change in Fear and Disgust Rating from pre- to posttreatment (across one week from pretreatment to posttreatment)
  Self-developed, computerized fear and disgust ratings of 30 pictures of various animals (i.e., different mammals, insects, rodents, reptiles, birds). Participants have to rate their level of fear and disgust for each animal separately on a scale from 0 to 100. Higher scores indicate greater fear and disgust for each animal.

CONTACTS AND LOCATIONS:
Overall Officials: Armin Zlomuzica, PhD, Principal Investigator — Ruhr-University Bochum
Locations (1):
- Mental Health Research and Treatment Center, Bochum, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Preusser F, Margraf J, Zlomuzica A. Generalization of Extinguished Fear to Untreated Fear Stimuli after Exposure. Neuropsychopharmacology. 2017 Dec;42(13):2545-2552. doi: 10.1038/npp.2017.119. Epub 2017 Jun 7. PMID 28589965
- [Background] Margraf, J. & Cwik, J. C. (2017). Mini-DIPS Open Access: Diagnostic Short-Interview for Mental Disorders. [Mini-DIPS Open Access: Diagnostisches Kurzinterview bei psychischen Störungen]. Bochum: Forschungs- und Behandlungszentrum für psychische Gesundheit, Ruhr-Universität. doi:10.13154/rub.102.9